CLINICAL TRIAL: NCT00406263
Title: Comparison of Scheimpflug Photos of the Crystalline Lens in Patients Who Have Undergone Vitrectony Surgery and Controls
Brief Title: Comparison of Scheimpflug Photos of the Crystalline Lens in Patients Who Have Undergone Vitrectomy Surgery and Controls
Status: Completed | Type: Observational
Sponsor: Barnes Retina Institute (Other)
Responsible Party: Principal Investigator, Rhonda Weeks, Nancy Holekamp, MD, Principal Investigator, Barnes Retina Institute
Other Study IDs: 06-1016
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Nuclear Sclerotic Cataract
Keywords: nuclear sclerotic cataract; cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Scheimpflug crystalline lens photographs — scheimpflug photographs

SUMMARY:
Progression of nuclear sclerotic cataract after pars plana vitrectomy has been recognized for many years The mechanism for the rapid progression of nuclear sclerotic cataract remains unclear. The objective of this trial is to evaluate and compare the level and progression of cataract advancement in controls versus eyes that have undergone 20-gauge pars plana vitrectomy and 25-gauge pars plana vitrectomy.

DETAILED DESCRIPTION:
Approximately 105 patients will be recruited to obtain 35 control eyes that have not had pars plana vitrectomy and 35 eyes who will have undergone 20-gauge pars plana vitrectomy and 35 eyes will have undergone 25-gauge pars plana vitrectomy. Scheimpflug crystalline lens photographs will be taken for evaluation of level and progression of cataract development.

ELIGIBILITY:
Inclusion Criteria:

* phakic eyes of patients that are scheduled to undergo pars plana vitrectomy,
* controls will be phakic eyes of patients that have not undergone andy kind of intraocular surgery,
* age 18 and older

Exclusion Criteria:

* any eye that is pseudophakic,
* has had previous vitreoretinal surgery,
* has had previous intravitreal injection,
* previous intraocular inflammatory condition such as uveitis,
* previous irradiation,
* any patient with a history of ocular malignancy,
* history of infectious intraocular condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing vitrectony surgery and controls
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2006-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Holekamp, MD, Principal Investigator — Barnes Retina Institute
Locations (1):
- Barnes Retina Institute, St Louis, Missouri, United States